CLINICAL TRIAL: NCT04265872
Title: Pilot Clinical Trial of Treatment With Bortezomib to Inhibit Homologous Recombination (HR) Followed by Pembrolizumab and Cisplatin in Patients With Chemotherapy-Pretreated Metastatic Triple Negative Breast Cancer
Brief Title: Bortezomib Followed by Pembrolizumab and Cisplatin in metTNBC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 020-008
Record Dates: First submitted 2020-01-23; First posted 2020-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib; pembrolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib followed by pembro/cis (Experimental): There is only one arm.
  Interventions: Drug: Bortezomib; pembrolizumab and cisplatin injections--bortezomib followed by pembro/cis

INTERVENTIONS:
Drug: Bortezomib; pembrolizumab and cisplatin injections--bortezomib followed by pembro/cis — injection into a vein
  Other Names: Keytruda, Velcade, Platinol

SUMMARY:
The hypothesis of this pilot trial is that administration of bortezomib will inhibit NHEJ in metastatic TNBC leading at the time of disease progression to metastases that are HR-deficient and sensitive to pembrolizumab and cisplatin therapy. The trial will include in depth analysis of the patients' TNBC genome and phosphoproteome to evaluate HR-proficiency and deficiency, and nuclear proteins that drive NHEJ, before and upon progression with bortezomib therapy.

DETAILED DESCRIPTION:
Seventy to 80% of breast cancers have a basal gene expression profile which is characterized by homologous recombination deficiency (HRD) and high proliferation. HRD leads to upregulation of the activity of the non-homologous end joining (NHEJ) error-prone pathway that repairs DNA double strand breaks, a process required for TNBC survival. The hypothesis of this pilot trial is that administration of bortezomib will inhibit NHEJ in metastatic TNBC leading at the time of disease progression to metastases that are HR-deficient and sensitive to pembrolizumab and cisplatin therapy. A patient with an exceptional complete and durable response of her primary-refractory metastatic TNBC with PI3K pathway inhibition followed at disease progression by nab paclitaxel/cisplatin provides the clinical rationale for the present trial which will utilize bortezomib to inhibit HR proficiency prior to administration of pembrolizumab and cisplatin in pretreated metastatic TNBC patients.

Patients will receive bortezomib until PD, followed by pembrolizumab and cisplatin until PD or a maximum of 6 cycles on study. If patients are responding, they may continue pembrolizumab at the physician's discretion off study. Metastatic TNBC patients will undergo core needle biopsies of a metastatic lesion at study entry and at disease progression from bortezomib for NGS, RPPA, and other molecular analyses.

Patients whose disease does not respond to pembrolizumab and cisplatin may be treated with standard of care breast cancer therapies off study, at the recommendation of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study if she meets all of the following criteria:

  1. Female patients ≥18 years of age
  2. Have a diagnosis of metastatic TNBC previously treated with standard anthracycline, cyclophosphamide, and taxane chemotherapy, unless there was a contraindication to doxorubicin, in which case prior treatment with this agent is not required. NOTE: TNBC defined as ER-negative tumors with < or = 10% tumor nuclei immunoreactivity, or "ER Low Positive" as defined by the updated ASCO/CAP guidelines 2020.
  3. Have not received more than 3 prior chemotherapy regimens for metastatic disease. Prior platinum and/or taxane therapy in the adjuvant or metastatic setting is permitted.
  4. Have locoregional (eg, breast, chest wall, regional lymphatic) or pulmonary or hepatic metastatic disease that is amenable to core needle biopsy. If a research biopsy from a patient's metastatic disease cannot be safely obtained, a skin biopsy is permitted. If a skin biopsy cannot be safely obtained, patients may still be eligible, per physician discretion.
  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (See Appendix I)
  6. Have adequate hematologic function, defined by:

     1. Absolute neutrophil count (ANC) >1500/μL
     2. Platelet count ≥100,000/μL
     3. Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
  7. Have adequate liver function, defined by:

     1. AST and ALT ≤2.5 x the upper limit of normal (ULN) or ≤5 x ULN in presence of liver metastases
     2. Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN
  8. Have adequate renal function, defined by:

     a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥30 mL/min
  9. Have adequate coagulation function, defined by:

     1. International Normalized Ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN.
     2. If patient is receiving anticoagulant therapy, PT or aPTT must be within therapeutic range of intended use of anticoagulants.
  10. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

      1. Brain metastases which have been treated
      2. Off-treatment with steroids for 2 weeks before administration of the first dose of bortezomib
      3. No ongoing requirement for dexamethasone or anti-epileptic drugs
      4. No clinical or radiological evidence of progression of brain metastases
  11. Patient must be accessible for treatment and follow-up.
  12. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* EXCLUSION CRITERIA

A patient will be ineligible for inclusion in this study if she meets any of the following criteria:

1. Has received a live vaccine within 30 days of the first dose of study treatment. NOTE: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (ie, FluMist ®) are live attenuated vaccines, and are not allowed.
2. Has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic therapy.
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
4. Has a known history of Human Immunodeficiency Virus (HIV)
5. Has known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
6. Has a history of non-infectious pneumonitis that required steroids or current pneumonitis
7. Has peripheral neuropathy ≥grade 2
8. Has completed previous radiotherapy for metastatic disease <2 weeks prior to study treatment initiation
9. Has an active infection requiring systemic therapy
10. Has significant cardiovascular disease, such as:

    1. History of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass grafting within the last 6 months
    2. Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV, or history of CHF NYHA class III or IV.
11. Has a known history of active tuberculosis
12. Women who are pregnant or lactating. All patients with reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug.
13. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

    1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
    2. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Treating Physician.
15. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study treatment (this would not include bortezomib while on study). Monoclonal antibody agents should have a 4-week (28 day) washout period.
16. Any other investigational or anti-cancer treatments while participating in this study
17. Any other active malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Calculate objective response rate (CR+PR) associated with bortezomib followed at disease progression with pembrolizumab and cisplatin in metastatic TNBC | 18 months
  objective response rate will be calculated by defining the proportion of patients who have a complete or partial response to the study therapy, as determined by the treating physician

SECONDARY OUTCOMES:
Calculate response | 18 months
  duration of response will be calculated from the time of tumor response to disease progression in patients responding to study therapy;

OTHER OUTCOMES:
evaluate research biopsy for homologous recombination deficiency via Next Generation Sequencing | 18 months
  research biopsies will be analyzed for homologous recombination deficiency via Next Generation Sequencing and Reverse Phase Protein Array

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — Texas Oncology
Locations (1):
- Baylor University Medical Center, Baylor Charles A Sammons Cancer Center, Dallas, Texas, United States